CLINICAL TRIAL: NCT00734201
Title: A Double-blind, Placebo-controlled, Parallel Group Study of the Effect of V24343 on Blood Pressure and Weight in Obese Subjects
Brief Title: Safety and Efficacy of Low Doses of V24343 in Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vernalis (R&D) Ltd (Industry)
Responsible Party: Steve Warrington, Medical Director, Hammersmith Medicines Research,
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: V24343-1Ob-03
Record Dates: First submitted 2008-08-06; First posted 2008-08-14 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Obesity
Keywords: Study effects on blood pressure and weight in obese subjects
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Randomised to a parallel group comparison of either one of four doses of study drug (1mg, 2mg, 5mg, 25mg) or placebo. Dosed once daily for 28 days
  Interventions: Drug: V24343

INTERVENTIONS:
Drug: V24343 — Oral, 1mg, 2 mg, 5 mg or 25 mg, or placebo, once daily for 28 days

SUMMARY:
Randomised, double-blind, parallel group comparison of four dose levels of V24343 and placebo to study the effect of V24343 on blood pressure and weight in obese subjects.

The primary variables, change in blood pressure (BP) and pulse, will be assessed both by outpatient ambulatory monitoring of vital signs and by regular clinic monitoring.

The efficacy of V24343 will be assessed by measurement of body weight, waist circumference, bioimpedance assessment of body composition and blood glucose.

Assay of plasma concentration of V24343 in blood samples collected at intervals after dosing will be used to assess the pharmacokinetics of V24343.

Other safety assessments comprise routine monitoring of adverse events; concomitant medication; clinical laboratory safety tests, 12-lead electrocardiograms (ECG) and self-completed psychiatric assessments.

ELIGIBILITY:
Inclusion Criteria: Subjects must:

* be healthy male subjects aged 18 to 60 years
* have a body mass index greater than or equal to 27 kg/m2
* have a waist measurement >94 cm
* have blood pressure (BP) within the ranges systolic BP (SBP): 90-150 mmHg; diastolic BP (DBP): 40-90 mmHg, based on mean of day time readings recorded during a 24 hour period of ambulatory monitoring:
* be willing to use an effective method of contraception (condom with a spermicidal contraceptive, or sterilised) for the duration of the study and for 3 months after the last dose of study medication
* have an acceptable medical and social history in the 12 months prior to screening
* be able to comply with the requirements of the entire study
* give written informed consent

Exclusion Criteria: Subjects must not:

* have received V24343 previously
* suffer from or have a history of anxiety or depression; have abnormal results on Patient Health Questionnaire 9 or Profile of Mood States (see Section 6.3.4.5)
* have a history of seizures (excluding febrile convulsions below 3 years of age)
* be male subjects whose female partners are trying to become pregnant within 3 months after the last dose of study medication
* have a significant medical condition or a history of such a condition that the Investigator considers should exclude the subject from the study
* have multiple drug allergies or be allergic to any of the components of V24343 study medication
* be smokers whom smoke more than 10 cigarettes per day
* consume more than 28 units of alcohol per week, or have a significant history of alcohol abuse
* have a positive test for alcohol or drugs of abuse at screening or admission to any of the treatment periods
* have donated blood or plasma in excess of 500 mL within 3 months of screening
* have been exposed to any new investigational agent within 3 months prior to study drug administration
* have clinically significant abnormalities on laboratory screening tests, particularly liver function and renal function tests (see Section 6.3.4.2)
* have clinically relevant abnormal physical findings on examination
* have clinically relevant abnormal findings on 12-lead ECG including a mean QTcB at screening ≥430 msec
* be seropositive for hepatitis B, hepatitis C or human immunodeficiency (HIV) viruses at screening
* have any medical or social reasons for not participating in the study raised by their General Practitioner/primary care physician
* have any other condition that might increase the risk to the individual or decrease the chance of obtaining satisfactory data, as assessed by the Investigator
* have had treatment with any prescription medicine within one month of first dose or any over-the-counter medicines, except for paracetamol, within one week of the first dose

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To examine any effects of V24343 on pulse and blood pressure (vital signs) | 24-hour on screening and pre-dose on Days 2, 26 and 56. Semi -recumbent and stand SBP , DBP and pulse, in duplicate at each time point.

SECONDARY OUTCOMES:
To determine if there is adequate differentiation between doses of V24343 associated with any effect on vital signs and those associated with efficacy (weight loss). | Body weight and wasit circumference: screen and time-matched to pre-dose on Days -1, 8, 15, 22, 29, 35, 42, 49 and 56.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Warrington, Principal Investigator — Medical Director
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom